CLINICAL TRIAL: NCT03264391
Title: Evaluation of Macular Vascular Changes in Behcet's Disease Using Optical Coherence Tomography Angiography
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menatallah Saleh, Principal Investigator, Assiut University
Other Study IDs: 17100296
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-05

CONDITIONS: Retinal Vasculitis; Behcet Syndrome
Keywords: OCT-A; Retinal vasculitis; Behcet's disease
MeSH Terms: conditions — Retinal Vasculitis; Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Behcet's disease is an important cause of retinal vasculitis and vision loss in Egypt. Fluorescein angiography is the standard method of diagnosis of retinal vasculitis. OCT angiography (OCT-A) is a recently developed method that can be used in the evaluation of retinal circulation. In this study, we will test the utility of OCT-A in diagnosis and follow up of retinal vascular changes in cases diagnosed with Behcet's disease that visit the outpatient uveitis clinic of Assiut University hospital, a major tertiary center in southern Egypt, over a one year duration. Also, correlation of OCT-A changes with visual acuity and hence prognosis will be described.

DETAILED DESCRIPTION:
Aim of the research To describe macular retinal vascular changes in patient with retinal vasculitis secondary to Behcet's disease both qualitatively and quantitatively.

Research design Type of the study: cross sectional analytical study Study Setting: Assuit University Hospital (Ophthalmology Department)

Study subjects:

1. Inclusion criteria:

   • Patients diagnosed with Behcet's disease with or without active uveitis
2. Exclusion criteria:

   * Patients less than 18 years old
   * Hazy media precluding clear fundus view.
   * Patients with very poor fixation.
3. Sample Size Calculation:

We will aim at recruiting all patients diagnosed with Behcet's disease in outpatient clinic who will meet the inclusion criteria within one year from the start of our project.

Methods Subject recruitment and obtaining consent Study subjects (Behcet's patients) will be recruited from patients attending uveitis and retina clinic of the ophthalmology Department, Faculty of Medicine, Assiut University. Written informed consent form will be obtained from each patient.

Baseline evaluation:

1. Full ocular examination including slit lamp and dilated fundus examinations. Also, measurement of the best corrected visual acuity (BCVA) using Snellen's chart will be done.
2. Thorough clinical history and review of other systems involvement as well as full drug history including use of topical and systemic medications.
3. Retinal vasculitis will be diagnosed by fundus examination. Additionally, fluorescein angiography may be done according to the discretion of the investigators to confirm the diagnosis.

Optical coherence tomography angiography imaging OCT imaging will be performed after pupillary dilatation using Topcon DRI OCT Triton platform which utilizes invisible 1050 nm light and obtains images at a speed of 100,000 A scans/sec.

First, B scans of the macula will be obtained and anatomical alterations of retinal architecture will be noted. Next, OCT angiography scans in a 4.5x 4.5 mm circle centered on the fovea will be then obtained. Analysis and interpretation of the enface images of the superficial and deep retinal capillary plexus as well as choriocapillaries will be performed. Areas of capillary dropout, abnormalities of retinal capillaries and vessels such as looping, dilated segments, microaneurysms as well as FAZ area will be documented.

Research outcome measures:

A. Primary (main):

1- Qualitative description of the retinal capillary plexus changes in the macular area

B. Secondary:

1. Quantification of the extent of macular ischemia by measuring the area of foveal avascular zone (FAZ).
2. Correlation between extent of macular vascular changes and visual acuity

Data management and analysis:

Data collection data will be recorded in the form of excel spreadsheets Computer software SPSS and Prism graphpad Statistical tests chi square test and Pearson correlation coefficient

ELIGIBILITY:
Inclusion Criteria:

* • Patients diagnosed with Behcet's disease

Exclusion Criteria:

* • Patients less than 18 years old

  * Hazy media precluding clear fundus view.
  * Patients with very poor fixation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Behcet's disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Qualitative description of the retinal capillary plexus changes in the macular area | 1 year

SECONDARY OUTCOMES:
Correlation between extent of macular vascular changes and visual acuity | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bazvand F, Zarei M, Ebrahimiadib N, Karkhaneh R, Davoudi S, Soleimanzadeh M, Sharifian E, Roohipoor R, Modjtahedi BS. Ocular Manifestations, Conventional Fundus Fluorescein Angiographic Findings, and Relationship Between Angiographic Findings and Visual Acuity in Behcet's Disease. Semin Ophthalmol. 2017;32(6):764-771. doi: 10.1080/08820538.2016.1178310. Epub 2016 Aug 10. PMID 27715380
- [Background] Fingler J, Readhead C, Schwartz DM, Fraser SE. Phase-contrast OCT imaging of transverse flows in the mouse retina and choroid. Invest Ophthalmol Vis Sci. 2008 Nov;49(11):5055-9. doi: 10.1167/iovs.07-1627. Epub 2008 Jun 19. PMID 18566457
- [Background] Leitgeb RA, Schmetterer L, Hitzenberger CK, Fercher AF, Berisha F, Wojtkowski M, Bajraszewski T. Real-time measurement of in vitro flow by Fourier-domain color Doppler optical coherence tomography. Opt Lett. 2004 Jan 15;29(2):171-3. doi: 10.1364/ol.29.000171. PMID 14744000
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Ocular+Manifestations%2C+Conventional+Fundus+Fluorescein+Angiographic+Findings%2C+and+Relationship+between+Angiographic+Findings+and+Visual+Acuity+in+Beh%C3%A7et%E2%80%99s+Disease
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Phase-contrast+OCT+imaging+of+transverse+flows+in+the+mouse+retina+and+choroid
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Real-time++measurement+of+in+vitro+flow+by+Fourier-domain+color+Doppler+optical+coherence+tomography.